CLINICAL TRIAL: NCT02343432
Title: Is the Efficacy of Epidural Steroid Injections Related to the Different Volume Injections? :A Randomised, Clinical Trial
Brief Title: Is the Efficacy of Epidural Steroid Injections Related to the Different Volume Injections?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neslihan Uztüre (Other)
Collaborators: University of Gaziantep (Other)
Responsible Party: Sponsor-Investigator, Neslihan Uztüre, assistant proffessor, Yeditepe University Hospital
Organization: Yeditepe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 03-2008/23
Record Dates: First submitted 2014-11-08; First posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Pain
Keywords: Anesthesia; Adverse Effect; Spinal; Epidural
MeSH Terms: conditions — Pain | interventions — Triamcinolone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Epidural Volume 10mL (Experimental): Epidural Volume 10mL, Intervention: Drug: Triamcinolone 80 mg Intervention: Drug: Epidural Volume 10mL Intervention: Drug: Bupivacaine 12.5mg
  Interventions: Drug: Triamcinolone; Drug: Epidural Volume; Drug: Bupivacaine
- Epidural Volume 15mL (Experimental): Epidural Volume 15mL, Intervention: Drug: Triamcinolone 80 mg Intervention: Drug: Epidural Volume 15 mL Intervention: Drug: Bupivacaine 12.5mg
  Interventions: Drug: Triamcinolone; Drug: Epidural Volume; Drug: Bupivacaine
- Epidural Volume 20mL (Experimental): Epidural Volume 20mL, Intervention: Drug: Triamcinolone 80 mg Intervention: Drug: Epidural Volume 20 mL Intervention: Drug: Bupivacaine 12.5mg
  Interventions: Drug: Triamcinolone; Drug: Epidural Volume; Drug: Bupivacaine

INTERVENTIONS:
Drug: Triamcinolone — Triamcinolone
  Other Names: Kelanocort
Drug: Epidural Volume — Epidural Volume
Drug: Bupivacaine — Bupivacaine
  Other Names: Marcaine

SUMMARY:
This study was aimed to investigate the impact of using different epidural volumes.

Patients with acute discogenic pain were included in the study.

DETAILED DESCRIPTION:
Objectives: This study was aimed to investigate the impact of using different epidural volumes.

Methods: Seventy five patients with acute discogenic pain were included in the study.The patients were randomly assigned to three groups. All patients received a single epidural dose of triamcinolone [80 mg] and 12.5 mg bupivacaine combination. The patients in Group 1, Group 2 and Group 3 received a volume of 10 mL, 15 mL, and 20 mL by epidural injections, respectively. The efficacy of treatment was assessed with VAS (visual analog scale) [O= no pain, 10 = unbearable pain], SLET(straight leg elevation test) [0° = worst, 85° = best], and Oswestry Disability Index; ODI [0% to 20%:minimal disability , 80% to 100%:bed bound patients] before and 2 weeks after the EPSI.

ELIGIBILITY:
Inclusion Criteria:

* acute discogenic pain with less than three months duration not responding to other modalities of conservative management [NSAIDs, physiotherapy, bracing, etc.],
* radiological disc bulging accompanying unilateral root impingement symptoms,
* an Oswestry daily activity score more than 20 percent, and
* resistance to treatment.

Exclusion Criteria:

* Patients with bilateral root impingement symptoms, neurological deficits, and/or history of previous lumbar disc surgery, severe cardiac, pulmonary, gastrointestinal, renal diseases, glaucoma, urinary retention, and/or known allergy to the drugs used in the study were excluded from the study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
VAS (visual analog scale) [O= no pain, 10 = unbearable pain] | 2 weeks
SLET(straight leg elevation test) [0° = worst, 85° = best] | 2 weeks
Oswestry Disability Index; ODI [0% to 20%:minimal disability , 80% to 100%:bed bound patients] | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye Budak, Study Director — University of Gaziantep

REFERENCES:
- [Background] Runu R, Sinha NK, Pai R, Shankar PR, Vijayabhaskar P. Our experience with epidural steroid injections in management of low backpain and sciatica. Kathmandu Univ Med J (KUMJ). 2005 Oct-Dec;3(4):349-54. PMID 16449834